CLINICAL TRIAL: NCT02122952
Title: Phase I Gene Transfer Clinical Trial for Spinal Muscular Atrophy Type 1 Delivering AVXS-101
Brief Title: Gene Transfer Clinical Trial for Spinal Muscular Atrophy Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-101; COAV101A12101 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Spinal Muscular Atrophy 1
Keywords: Gene Transfer; Gene Therapy; Adeno-associated virus; Survival Motor Neuron; SMN; AAV9
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 6.7 X 10^13 vg/kg of AVXS-101 delivered one-time through a venous catheter inserted into a peripheral vein (n=3)
  Interventions: Biological: AVXS-101
- Cohort 2 (Experimental): 2.0 X 10^14 vg/kg of AVXS-101 delivered one-time through a venous catheter inserted into a peripheral vein (n=12)
  Interventions: Biological: AVXS-101

INTERVENTIONS:
Biological: AVXS-101 — Self-complementary AAV9 carrying the SMN gene under the control of a hybrid CMV enhancer/chicken-β-actin promoter
  Other Names: Zolgensma

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of intravenous delivery of AVXS-101 as a treatment of spinal muscular atrophy Type 1 (SMN1).

DETAILED DESCRIPTION:
The study will evaluate safety and efficacy of gene therapy in spinal muscular atrophy Type 1 (SMA1) patients. SMA is caused by low levels of the survival motor neuron (SMN) protein, and affects all muscles in the body. There is no effective treatment for SMA and current drug therapy has been unsuccessful in stabilizing or reversing this disease. Only supportive care is currently possible.

Open-label, dose-escalation clinical trial of AVXS-101 injected intravenously through a peripheral limb vein. Short-term safety will be evaluated over a two year period. Patients will be tested at baseline and return for follow up visits on days 7, 14, 21, 30, followed by once every month through 12 months post dose, and then every three months through two (2) years post infusion. Unscheduled visits may occur if the PI determines that they are necessary.

The primary analysis for efficacy will be assessed when all patients reach 13.6 months of age (a database lock will be performed at the time point at which all patients reach 13.6 months of age). A follow-up safety analysis will be completed at the time point at which the last patient reaches 24 months post-dose.

Upon completion of the 2-year study period, patients will be monitored annually as per standard of care for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Six or nine months of age and younger (depending on cohort) on day of vector infusion with Type 1 SMA as defined by the following features:

  * Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 2 copies of SMN2.
  * Onset of disease at birth up to 6 months of age.
  * Hypotonia by clinical evaluation with delay in motor skills, poor head control, round shoulder posture and hypermobility of joints.

Exclusion Criteria:

* Active viral infection (includes HIV or serology positive for hepatitis B or C)
* Use of invasive ventilatory support (tracheotomy with positive pressure)* or pulse oximetry <95% saturation.
* Patients may be put on non-invasive ventilator support (BiPAP) for less than 16 hours a day at the discretion of their physician or research staff.
* Concomitant illness that in the opinion of the PI creates unnecessary risks for gene transfer
* Concomitant use of any of the following drugs: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (e.g. corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab)
* Patients with Anti-AAV9 antibody titers >1:50 as determined by ELISA binding immunoassay.
* Abnormal laboratory values considered clinically significant (GGT > 3XULN, bilirubin ≥ 3.0 mg/dL , creatinine ≥ 1.8 mg/dL, Hgb < 8 or > 18 g/Dl; WBC > 20,000 per cmm) Participation in a recent SMA treatment clinical trial that in the opinion of the PI creates unnecessary risks for gene transfer.
* Family does not want to disclose patient's study participation with primary care physician and other medical providers.
* Patient with signs of aspiration based on a swallowing test and unwilling to use an alternative method to oral feeding.
* Patients with a single base substitution in SMN2 (c.859G>C in exon 7) will be excluded based on predicted mild phenotype.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Bevan AK, Duque S, Foust KD, Morales PR, Braun L, Schmelzer L, Chan CM, McCrate M, Chicoine LG, Coley BD, Porensky PN, Kolb SJ, Mendell JR, Burghes AH, Kaspar BK. Systemic gene delivery in large species for targeting spinal cord, brain, and peripheral tissues for pediatric disorders. Mol Ther. 2011 Nov;19(11):1971-80. doi: 10.1038/mt.2011.157. Epub 2011 Aug 2. PMID 21811247
- [Background] Bevan AK, Hutchinson KR, Foust KD, Braun L, McGovern VL, Schmelzer L, Ward JG, Petruska JC, Lucchesi PA, Burghes AH, Kaspar BK. Early heart failure in the SMNDelta7 model of spinal muscular atrophy and correction by postnatal scAAV9-SMN delivery. Hum Mol Genet. 2010 Oct 15;19(20):3895-905. doi: 10.1093/hmg/ddq300. Epub 2010 Jul 16. PMID 20639395
- [Background] Foust KD, Wang X, McGovern VL, Braun L, Bevan AK, Haidet AM, Le TT, Morales PR, Rich MM, Burghes AH, Kaspar BK. Rescue of the spinal muscular atrophy phenotype in a mouse model by early postnatal delivery of SMN. Nat Biotechnol. 2010 Mar;28(3):271-4. doi: 10.1038/nbt.1610. Epub 2010 Feb 28. PMID 20190738 (Retraction: PMID 36203015 Nat Biotechnol. 2022 Nov;40(11):1692)
- [Background] Foust KD, Nurre E, Montgomery CL, Hernandez A, Chan CM, Kaspar BK. Intravascular AAV9 preferentially targets neonatal neurons and adult astrocytes. Nat Biotechnol. 2009 Jan;27(1):59-65. doi: 10.1038/nbt.1515. Epub 2008 Dec 21. PMID 19098898
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- [Derived] Lowes LP, Alfano LN, Arnold WD, Shell R, Prior TW, McColly M, Lehman KJ, Church K, Sproule DM, Nagendran S, Menier M, Feltner DE, Wells C, Kissel JT, Al-Zaidy S, Mendell J. Impact of Age and Motor Function in a Phase 1/2A Study of Infants With SMA Type 1 Receiving Single-Dose Gene Replacement Therapy. Pediatr Neurol. 2019 Sep;98:39-45. doi: 10.1016/j.pediatrneurol.2019.05.005. Epub 2019 May 13. PMID 31277975
- [Derived] Dabbous O, Maru B, Jansen JP, Lorenzi M, Cloutier M, Guerin A, Pivneva I, Wu EQ, Arjunji R, Feltner D, Sproule DM. Survival, Motor Function, and Motor Milestones: Comparison of AVXS-101 Relative to Nusinersen for the Treatment of Infants with Spinal Muscular Atrophy Type 1. Adv Ther. 2019 May;36(5):1164-1176. doi: 10.1007/s12325-019-00923-8. Epub 2019 Mar 16. PMID 30879249
- [Derived] Al-Zaidy S, Pickard AS, Kotha K, Alfano LN, Lowes L, Paul G, Church K, Lehman K, Sproule DM, Dabbous O, Maru B, Berry K, Arnold WD, Kissel JT, Mendell JR, Shell R. Health outcomes in spinal muscular atrophy type 1 following AVXS-101 gene replacement therapy. Pediatr Pulmonol. 2019 Feb;54(2):179-185. doi: 10.1002/ppul.24203. Epub 2018 Dec 12. PMID 30548438
- [Derived] Mendell JR, Al-Zaidy S, Shell R, Arnold WD, Rodino-Klapac LR, Prior TW, Lowes L, Alfano L, Berry K, Church K, Kissel JT, Nagendran S, L'Italien J, Sproule DM, Wells C, Cardenas JA, Heitzer MD, Kaspar A, Corcoran S, Braun L, Likhite S, Miranda C, Meyer K, Foust KD, Burghes AHM, Kaspar BK. Single-Dose Gene-Replacement Therapy for Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1713-1722. doi: 10.1056/NEJMoa1706198. PMID 29091557
- See also: Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy
- See also: AveXis, Inc — http://avexis.com/
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period May 2014 - Dec 2015
Pre-assignment Details: 30 day screening period prior to enrollment and dosing.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 3 | 12
Completed | 3 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 12 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.33 (0.751) | 3.42 (2.063) | 4.00 (2.209)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 10 | 13
  Hispanic or Latino | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 15
SMN2 copy number = 2 [Count of Participants; unit: Participants] | 3 | 12 | 15
bi-allelic deletions of SMN1 [Count of Participants; unit: Participants] | 3 | 12 | 15
Exon 7 gene modifier mutation [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced One Grade III or Higher Unanticipated, Treatment-related Toxicity That Presents With Clinical Symptoms and Requires Medical Treatment
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 12
Participants | 1 | 3

2. Secondary Outcome: Number of Participants Who Experienced Permanent Ventilation or Death
Description: Permanent ventilation was defined as the requirement of ≥ 16-hour respiratory assistance, including non-invasive ventilatory support, per day continuously for ≥ 2 weeks in the absence of an acute reversible illness, excluding perioperative ventilation.
Time Frame: Up to 13.6 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 12
Participants | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in Mean Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) Score
Description: Score ranges from 0 to 64, where 64 is the maximum possible score. A higher score is indicative of higher/better motor function. CHOP-INTEND assessments were discontinued once patients achieved higher functioning status, so the number of available data points decreased over time.
Time Frame: Baseline to 24 months post-dose
Population: Includes all treated participants with non-missing data. For a major, systemic, and externally imposed limitation of movement that prevented accurate assessment of multiple items, the total score was regarded as missing. Also, CHOP-INTEND assessments were discontinued once participants achieved higher functioning status (2 consecutive scores ≥62).
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 6
Percentage Change |  | 30.7 (145.61)

4. Secondary Outcome: Number of Participants With Assessed Improvement in Motor Function
Description: Improvement in motor function was determined by achievement of developmental milestones, specifically achievement of ability to sit unassisted for at least 30 seconds, determined by physical therapist and confirmed by an independent central video reviewer. Achievement of functional independent sitting was defined as the ability to maintain a sitting position independently for at least 30 seconds as confirmed per video evaluation by an expert central reviewer based on videos taken either at scheduled visits or provided by the parent/legal guardian.
Time Frame: 24 months post-dose
Population: full analysis set- all treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 12
Participants | 0 | 9
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Data for the current study were compared to historical control data (Pediatric Neuromuscular Clinical Research [PNCR], Finkel et al 2014 - PubMed 25080519) where 0 participants were able to sit independently; Test type: Superiority; p < 0.001, One-sided Exact Binomial Test

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the single dose of study treatment until 24 months post dose
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/3 | 10/12
Other Adverse Events (participants affected / at risk) | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=12)
pneumonia (Infections and infestations) | 0 (0) | 7 (10)
rhinovirus infection (Infections and infestations) | 0 (0) | 2 (5)
enterovirus infection (Infections and infestations) | 0 (0) | 2 (3)
parainfluenzae virus infection (Infections and infestations) | 1 (1) | 2 (2)
respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
adenovirus infection (Infections and infestations) | 0 (0) | 2 (2)
human rhinovirus test positive (Investigations) | 0 (0) | 2 (2)
lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
penumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (2)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
transaminases increased (Investigations) | 1 (1) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
enterovirus test positive (Investigations) | 0 (0) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
norovirus test positive (Investigations) | 0 (0) | 1 (1)
oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=12)
constipation (Gastrointestinal disorders) | 1 (1) | 6 (8)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (6)
vomiting (Gastrointestinal disorders) | 0 (0) | 8 (11)
pyrexia (General disorders) | 1 (1) | 7 (12)
bronchiolitis (Infections and infestations) | 0 (0) | 3 (3)
conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
ear infection (Infections and infestations) | 1 (1) | 2 (2)
enterovirus infection (Infections and infestations) | 1 (1) | 3 (4)
gastroenteritis viral (Infections and infestations) | 0 (0) | 5 (5)
otitis media (Infections and infestations) | 2 (6) | 2 (3)
parainfluenzae virus infection (Infections and infestations) | 0 (0) | 2 (2)
pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2)
pneumonia (Infections and infestations) | 0 (0) | 4 (4)
rhinovirus infection (Infections and infestations) | 1 (1) | 4 (5)
upper respiratory tract infection (Infections and infestations) | 1 (3) | 9 (25)
urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
human rhinovirus test positive (Investigations) | 0 (0) | 3 (4)
transaminases increased (Investigations) | 0 (0) | 2 (2)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (11)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (9)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
food allergy (Immune system disorders) | 0 (0) | 1 (1)
hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
catheter site inflammation (General disorders) | 1 (1) | 0 (0)
catheter site pain (General disorders) | 0 (0) | 1 (1)
pain (General disorders) | 0 (0) | 1 (1)
secretion discharge (General disorders) | 0 (0) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
enterovirus test positive (Investigations) | 0 (0) | 1 (1)
eosinophil count increased (Investigations) | 0 (0) | 1 (1)
haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
blepharitis (Eye disorders) | 0 (0) | 1 (2)
chalazion (Eye disorders) | 1 (1) | 0 (0)
dry eye (Eye disorders) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
mastication disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
hyperglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 0 (0) | 1 (1)
lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
otitis externa (Infections and infestations) | 0 (0) | 1 (1)
otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
viral infection (Infections and infestations) | 0 (0) | 1 (1)
wound infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Link to the full study results: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17849

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will provide proposed publication or presentation for review 60 days prior; Sponsor informs PI in writing of revisions required to protect Sponsor's confidential and proprietary technical information and to address inaccurate data or inappropriate interpretations. At expiration of such 60 days, PI may proceed unless Sponsor has notified in writing that such proposed publication or presentation discloses the Sponsor's confidential and proprietary technical information.

DOCUMENTS (2):
  • Study Protocol (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT02122952/Prot_001.pdf
  • Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02122952/SAP_000.pdf